CLINICAL TRIAL: NCT00632086
Title: A Phase 1, Open-Label, Randomized, 3-Way Crossover Study to Evaluate the Relative Bioavailability of a Single Oral Dose of Aspirin Administered as PA32540 (Aspirin/Omeprazole) or as the Aspirin Component of PA32540 or as Ecotrin® 325 mg in Healthy Volunteers
Brief Title: Evaluate Relative Bioavailability of PA32540 (Asa/Omeprazole), Its Aspirin Component, and Ecotrin® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Connie Powers, Pozen
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PA32540-104
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: PK
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Single oral dose of 325 mg aspirin administered as PA32540
  Interventions: Drug: PA32540
- 2 (Experimental): aspirin core
  Interventions: Drug: aspirin component of PA32540
- 3 (Active Comparator): active
  Interventions: Drug: Ecotrin

INTERVENTIONS:
Drug: PA32540
  Arms: 1
Drug: aspirin component of PA32540 — The 325 mg aspirin component of PA32540
  Arms: 2
Drug: Ecotrin — 325 mg Ecotrin
  Arms: 3

SUMMARY:
Study to determine a single dose bioavailablity of PA32540 is similar to EC aspirin 325 mg with respect to salicylic acid.

ELIGIBILITY:
Inclusion Criteria:

* Standard for PK
* Ages 18-55 years old
* Males and females

Exclusion Criteria:

* Standard for PK

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)